CLINICAL TRIAL: NCT01643915
Title: Behavior Management Using Audiovisual Tools in Pediatric Dental Patients
Brief Title: Behavior Management Using Audiovisual Tools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Francisco Guinot-Jimeno, DDS, MsC, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: UIC-ODP-2
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Disruptive Global Behavior During Previous Treatment Visits
Keywords: Audiovisual distraction; Pediatric dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (Active Comparator): Patients with conventional treatment. No distraction method during the treatment visits.
  Interventions: Behavioral: No distraction method
- Experimental group 1 (Experimental): Patients will see a cartoon film in a screen attached to the ceiling, just above the dental chair during the second treatment visit.
  Interventions: Behavioral: Distraction method
- Experimental group 2 (Experimental): Patients will see a cartoon film with with Rimax® multimedia eyeglasses that occlude the environment partially during the second treatment visit.
  Interventions: Behavioral: Distraction method

INTERVENTIONS:
Behavioral: No distraction method — Patients with conventional treatment. No distraction method during the treatment visits.
  Arms: Control group
Behavioral: Distraction method — Patients will see a cartoon film in a screen attached to the ceiling, just above the dental chair during the second treatment visit.
  Arms: Experimental group 1
Behavioral: Distraction method — Patients will see a cartoon film with with Rimax® multimedia eyeglasses that occlude the environment partially during the second treatment visit.
  Arms: Experimental group 2

SUMMARY:
The aim of the study was to assess whether the behavior, anxiety, and pain of pediatric patients during dental treatment improves when a cartoon film is viewed or a videogame is played as methods of distraction.

DETAILED DESCRIPTION:
Each patient required a minimum of 2 visits for restorative treatment in a mandibular quadrant and had undergone a previous restorative dental experience. All parents or guardians of the children who participated in the study were informed about the study before enrolment, and gave their voluntary consent. Each visit lasted approximately 35 minutes and involved restorative treatment in a mandibular quadrant with an alveolar nerve block. The parents were not present in the operating room during the treatment. The maximum time between the 2 treatment sessions was 2 weeks. Before the start of each treatment session, as a part of the standard process of a paediatric dental visit, the child was given an explanation as to what the visit would comprise, with the aim of interrupting the treatment as little as possible. The children knew at the beginning of the first appointment (control) that they would be able to watch a movie or play a videogame during their next visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4-9 years.
* Patients who required a minimum of 2 visits for restorative treatment.
* Patients who had previously shown disruptive behavior (Frankl Behavior Rating Scale 1 or 2) during dental restorative treatment or pulp therapy.

Exclusion Criteria:

* Patients with reduced audiovisual capabilities.
* Patients with psychological disorders.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Global behavior during the treatment | 14 days

SECONDARY OUTCOMES:
Parental perception of patients' anxiety | 14 days
Self-reported anxiety during the treatment | 14 days
Pain during the treatment | 14 days
Heart rate during the treatment measures in different time points | 14 days
Degree of acceptance of the distraction method by the pediatric patient | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

REFERENCES:
- [Background] Ram D, Shapira J, Holan G, Magora F, Cohen S, Davidovich E. Audiovisual video eyeglass distraction during dental treatment in children. Quintessence Int. 2010 Sep;41(8):673-679. PMID 20657857
- [Background] El-Sharkawi HF, El-Housseiny AA, Aly AM. Effectiveness of new distraction technique on pain associated with injection of local anesthesia for children. Pediatr Dent. 2012 Mar-Apr;34(2):e35-8. PMID 22583875